CLINICAL TRIAL: NCT04671888
Title: Chronic Obstructive Pulmonary Disease (COPD) Monitoring
Acronym: COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medtronic BRC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MDT19035
Record Dates: First submitted 2020-12-04; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: COPD; COPD Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COPD patients (Experimental)
  Interventions: Other: exercises

INTERVENTIONS:
Other: exercises — COPD patients will be asked to wear a data logger system to collect EMG data and respiration parameters during exercise that simulate daily activity (i.e., walking, cycling)

SUMMARY:
The present feasibility study aims at assessing whether the EMG of respiratory muscles can serve as an objective marker of dyspnea in COPD patients.

The study aims also at evaluating the changes in physiological parameters (i.e., EMG, respiration rate, heart rate, temperature, and SpO2) occurring when simulating daily activities before, during and after acute exacerbations. All this information can be useful to detect the exacerbations earlier or to provide better treatment during the exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a clinical diagnosis of COPD
* mMRC (Modified Medical Research Council) Dyspnea Scale Score > 1
* Subject must be indicated for regular inpatient pulmonary rehabilitation
* Subject must be hyperinflated, defined as residual volume (RV)>120% of the predicted value, measured by whole body plethysmography
* Subject must be willing to provide Informed Consent for their participation in the study
* Subject must be ≥18 years of age

Exclusion Criteria:

* Subjects who are unable/unwilling to voluntarily participate in the study
* Subjects who cannot read/write
* Subjects who are dependent on oxygen and/or unfit to wear a mask during sub- maximal constant work rate test (CWRT)
* Subject has congenital heart disease
* Subject has unstable coronary artery disease
* Subject has an active implanted cardiac device (i.e. IPG, ICD)
* Subject has heart failure NYHA 4
* Subject presents any concomitant condition which in the opinion of the investigator would not allow a safe participation in the study
* Subject is legally incompetent
* Subject is pregnant or has suspect to be pregnant
* Subject is enrolled in a concurrent study that may confound the results of this study without documented pre-approval from Medtronic study manager
* BORG scale assessment is evaluated as unreliable due to patient's cognitive condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Correlation between EMG and BORG scale during sub-maximal constant work rate test (CWRT) exercise | through study completion, an average of 3 months
  To evaluate the correlation between EMG amplitude collected by means of the data logger system and BORG scale during sub-maximal CWRT exercise.
Correlation between EMG and BORG scale during rehabilitation exercise | through study completion, an average of 3 months
  To evaluate the correlation between EMG amplitude collected by means of the data logger system and BORG scale during rehabilitation exercise .

SECONDARY OUTCOMES:
EMG (Exacerbation symptoms assessment) | through study completion, an average of 3 months
  To evaluate the change of EMG amplitude between stable condition and an acute exacerbation episode
Respiration rate (Exacerbation symptoms assessment) | through study completion, an average of 3 months
  To evaluate the change of respiration rate between stable condition and an acute exacerbation episode
Transcutaneous oxygen saturation (Exacerbation symptoms assessment) | through study completion, an average of 3 months
  To evaluate the change of transcutaneous oxygen saturation between stable condition and an acute exacerbation episode
BORG scale (Exacerbation symptoms assessment) | through study completion, an average of 3 months
  To evaluate the change of BORG scale between stable condition and an acute exacerbation episode
Correlation between respiration rate and BORG scale | through study completion, an average of 3 months
  To evaluate the correlation between the respiration rate and BORG scale
Correlation between transcutaneous oxygen saturation and BORG scale | through study completion, an average of 3 months
  To evaluate the correlation between transcutaneous oxygen saturation and BORG scale

CONTACTS AND LOCATIONS:
Overall Officials: Martijn Spruit, Principal Investigator — Center of Expertise for Chronic Organ Failure

IPD SHARING:
Plan to Share IPD: No